CLINICAL TRIAL: NCT05310825
Title: An Examination of the Effect on Various Factors of Bed Baths Applied by Two Different Methods in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Bursa Uludag University, Department of Nursing, Uludag University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/1-23
Record Dates: First submitted 2022-03-01; First posted 2022-04-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2022-03

CONDITIONS: Patient Care
Keywords: Intensive Care Patients; Bed Baths; nursing; hemodynamic factors; wipe bath

STUDY DESIGN:
Intervention Model Description: The research is planned as a randomized, controlled, crossover and experimental study
Masking Description: The intervention and measurements were carried out by the first researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry Wiping Bath with Single-Use Wipes (Experimental): Cleaning wipes will be used in the bathing process which do not contain alcohol, paraben or latex. Before taking them out of the packet, the wipes to be used in the bathing will be heated according to usage instructions at 850 W for 50 seconds in a microwave oven which will be brought by the researcher. After heating, the temperature of the cleaning towels will be measured with an infrared thermometer. The reason for heating the wipes is to bring them to the same temperature as the bath water and thus to prevent any factors arising from a temperature difference.
  Interventions: Other: Dry Wiping Bath with Single-Use Wipes
- Traditional Body Wiping Bath (Other): Before bathing, two basins will be filled with a suitable amount (2/3 of the basin) of water at a suitable temperature (43°C). Water temperature will be measured by the researcher with a water thermometer. This thermometer will be used to bring the bath water to the correct temperature. Neutral soap will be added to the water of one basin, while the water of the other basin will be used for rinsing. The neutral soap to be used will not dry the skin or cause chafing or irritation, and it will be noon-allergenic. At the same time, soap with these characteristics is one which is routinely used for patient hygiene in the intensive care unit where the study will be conducted. The rubbing cloth to be used with both the soapy and the rinsing water in the routine procedure will have an inner layer of pure cotton with an outer layer of hydrophilic gauze. The patient's body wash will be performed with this cloth, using foam from the soapy water.
  Interventions: Other: Traditional Body Wiping Bath

INTERVENTIONS:
Other: Dry Wiping Bath with Single-Use Wipes — Cleaning wipes will be used in the bathing process which do not contain alcohol, paraben or latex. These wipes are a product routinely used in patient hygiene procedures in the intensive care unit where the study is to be conducted. Before taking them out of the packet, the wipes to be used in the bathing will be heated according to usage instructions at 850W for 50 seconds in a microwave oven which will be brought by the researcher The steps to be followed in the wiping procedures of bath will be, in order, cleaning the patient's face area (the eyes will only be cleaned with rinsing water), the ears on each side, the arms, the hands, the breast and chest area, the legs on each side, the feet, the back, and finally, the perineum and anal area, after which the washing procedure will be terminated.
  Arms: Dry Wiping Bath with Single-Use Wipes
Other: Traditional Body Wiping Bath — The rubbing cloth to be used with both the soapy and the rinsing water in the routine procedure will have an inner layer of pure cotton with an outer layer of hydrophilic gauze. The patient's body wash will be performed with this cloth, using foam from the soapy water. As soon as the bathing procedure is commenced, a chronometer will be started by another nurse who is independent of the study.
  The steps to be followed in the wiping procedures of bath will be, in order, cleaning the patient's face area (the eyes will only be cleaned with rinsing water), the ears on each side, the arms, the hands, the breast and chest area, the legs on each side, the feet, the back, and finally, the perineum and anal area, after which the washing procedure will be terminated
  Arms: Traditional Body Wiping Bath

SUMMARY:
The aim of this study is to evaluate the effect on various hemodynamic factors (breathing, pulse, blood pressure, peripheral oxygen saturation) of patients in intensive care units and the time taken for the procedure of a traditional wiping bed bath performed with soap and water) and one performed with single-use wipes.

The research is planned as a randomized, controlled, crossover and experimental study. Because it is planned as a crossover study, patients will be in both the experimental and the control group. The research will be conducted in the General Surgery Intensive Care Unit of Bursa Uludağ University Health Applications Research Center, Turkey. The population of the study will consist of patients in the Intensive Care Unit.

Patients participating in the study will be given two types of wiping body bath. One of these will be a wiping body bath performed with soap and water, which is accepted as a traditional bed bath. The other will be a body wiping bath performed with single-use wipes, which is accepted as a dry bath. All bathing procedures in the study will be conducted by the same researcher.

During both types of bathing, an assistant patient care worker will help the researcher in the process of turning the patient. Before starting, this assistant will be given information on the steps in bed bathing by the researcher. Each patient will be given a traditional wiping bed bath and a dry wiping bath with single-use wipes. Because this is a crossover study, the patient will be part of both the experimental and the control group.

The patient's first bath will be within the first 24 hours of entry to the intensive care unit. The randomization of each patient's bathing will be carried out according to a randomization list created on a computer and the patients will be assigned to the study groups by the randomization method. In this way, patients will be assigned to group 1 (traditional body wipe bathing with soap and water) and group 2 (dry body wipe bathing with single-use wipes). The bathing order will be carried out according to the randomization for each patient, and in this way, the patient's first bath will be performed as dry body wipe bathing with single-use wipes or as traditional body wipe bathing with soap and water. For each bath, a minimum interval of 24 hours (washing) will be left to prevent one intervention from affecting the other.

Immediately before giving each type of bed bath, every five minutes during the bathing procedure, immediately after finishing the bathing procedure and 30 minutes after finishing the bathing procedure, the patient's pulse, blood pressure, body temperature, breathing rate and oxygen saturation will be measured by a different nurse, and the values obtained together with the time taken for the procedure will be entered on the Patient Bathing Monitoring Form.

The steps to be followed in the wiping procedures of both baths will be, in order, cleaning the patient's face area (the eyes will only be cleaned with rinsing water), the ears on each side, the arms, the hands, the breast and chest area, the legs on each side, the feet, the back, and finally, the perineum and anal area, after which the washing procedure will be terminated.

After bathing, the patient's bedsheets and clothing will be changed and waste will be removed from the area. If the bandaging in the patient's operation area has not yet been removed, the operation area will not be washed. Also, the chronometer will be stopped by a nurse who is independent of the study immediately after the bathing procedure is completed, and the time taken for the procedure will be entered on the form.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect on various hemodynamic factors (breathing, pulse, blood pressure, peripheral oxygen saturation) of patients in intensive care units and the time taken for the procedure of a traditional wiping bed bath performed with soap and water) and one performed with single-use wipes.

The research is planned as a randomized, controlled, crossover and experimental study. Because it is planned as a crossover study, patients will be in both the experimental and the control group. The research will be conducted in the General Surgery Intensive Care Unit of Bursa Uludağ University Health Applications Research Center. The population of the study will consist of patients in the Intensive Care Unit. The size of the study sample was statistically determined with the program G*Power 3.1.7. In the power analysis conducted to determine the sample size, the two bathing methods were compared, and the effect size of blood pressure and breathing rate was determined. For a significance level of 0.05 and 80% power, it was calculated that a total of 22 patients were needed.

Patients with serious burns and/or diarrhea, open wound bandaging or amputations of the upper or lower extremities, those whose blood pressure measurements cannot be taken because of plaster or for other reasons, those who are discharged or die during data collection, and those who do not agree to participate in the study will not be included in the research.

A Patient Description Form and a Patient Bathing Monitoring Form will be used to obtain data.

Patient Description Form: This from will have questions on patients' age, gender, marital status, education level, medical diagnosis, length of time in hospital and in intensive care, chronic illnesses if any are present, method of connection to ventilation, and sedation status.

Patient Bathing Monitoring Form: This form will be used before, during, immediately after and 30 minutes after bathing to record heart rate, blood pressure, body temperature, breathing rate, oxygen saturation values and the time taken for bathing.

Data Collection Intensive care patients will be included in the study who themselves agree to participate, or who are not in a condition to decide, but their legal next of kin voluntarily give their agreement.

Patients participating in the study will be given two types of wiping body bath. One of these will be a wiping body bath performed with soap and water, which is accepted as a traditional bed bath. The other will be a body wiping bath performed with single-use wipes, which is accepted as a dry bath. All bathing procedures in the study will be conducted by the same researcher.

Before both of the bed bath procedures, the environment will be adjusted to a temperature of 25°C and 55% airflow. In order to achieve this, there is a room thermometer in intensive care, showing airflow and environment temperature. Screens will be drawn around the patient's bed and the patient's privacy will be respected. The necessary precautions will be taken to ensure that the patient does not fall. Before bathing, the windows and door of the intensive care unit will be closed against any possible draughts in the room. The procedure to be used will be explained to the patients before bathing, using verbal and non-verbal communication techniques. Descriptive information of the patients who agree to participate in the study will be recorded on the Patient Description Form, taken either from themselves or from their files.

During both types of bathing, an assistant patient care worker will help the researcher in the process of turning the patient. Before starting, this assistant will be given information on the steps in bed bathing by the researcher. Each patient will be given a traditional wiping bed bath and a dry wiping bath with single-use wipes. Because this is a crossover study, the patient will be part of both the experimental and the control group The patient's first bath will be within the first 24 hours of entry to the intensive care unit. The randomization of each patient's bathing will be carried out according to a randomization list created on a computer, and the patients will be assigned to the study groups by the randomization method. In this way, patients will be assigned to group 1 (traditional body wipe bathing with soap and water) and group 2 (dry body wipe bathing with single-use wipes). The bathing order will be carried out according to the randomization for each patient, and in this way, the patient's first bath will be performed as dry body wipe bathing with single-use wipes or as traditional body wipe bathing with soap and water. For each bath, a minimum interval of 24 hours (washing) will be left to prevent one intervention from affecting the other.

Immediately before giving each type of bed bath, every five minutes during the bathing procedure, immediately after finishing the bathing procedure and 30 minutes after finishing the bathing procedure, the patient's pulse, blood pressure, body temperature, breathing rate and oxygen saturation will be measured by a different nurse, and the values obtained together with the time taken for the procedure will be entered on the Patient Bathing Monitoring Form.

The steps to be followed in the wiping procedures of both baths will be, in order, cleaning the patient's face area (the eyes will only be cleaned with rinsing water), the ears on each side, the arms, the hands, the breast and chest area, the legs on each side, the feet, the back, and finally, the perineum and anal area, after which the washing procedure will be terminated.

Traditional Body Wiping Bath Procedure: Before bathing, two basins will be filled with a suitable amount (2/3 of the basin) of water at a suitable temperature (43°C). Water temperature will be measured by the researcher with a water thermometer. This thermometer will be used to bring the bath water to the correct temperature. Neutral soap will be added to the water of one basin, while the water of the other basin will be used for rinsing. The neutral soap to be used will not dry the skin or cause chafing or irritation, and it will be noon-allergenic. At the same time, soap with these characteristics is one which is routinely used for patient hygiene in the intensive care unit where the study will be conducted. The rubbing cloth to be used with both the soapy and the rinsing water in the routine procedure will have an inner layer of pure cotton with an outer layer of hydrophilic gauze. The patient's body wash will be performed with this cloth, using foam from the soapy water. As soon as the bathing procedure is commenced, a chronometer will be started by another nurse who is independent of the study.

After the procedure of washing with foam, the patient's whole body will be wiped with rinsing water. After this is completed, the patient's body will be dried with their own personal towel. In wiping each area, a different rubbing cloth will be used. Afterwards, the patient's bedsheets and clothing will be changed and waste will be removed from the area. If the bandaging in the patient's operation area has not yet been removed, the operation area will not be washed. Also, the chronometer will be stopped by a nurse who is independent of the study immediately after the bathing procedure is completed, and the time taken for the procedure will be entered on the form.

Dry Wiping Bath with Single-Use Wipes: Cleaning wipes will be used in the bathing process which do not contain alcohol, paraben or latex. These wipes are a product routinely used in patient hygiene procedures in the intensive care unit where the study is to be conducted. Before taking them out of the packet, the wipes to be used in the bathing will be heated according to usage instructions at 850W for 50 seconds in a microwave oven which will be brought by the researcher. After heating, the temperature of the cleaning towels will be measured with an infrared thermometer. It is aimed that the temperature should be approximately 43 degrees. The reason for heating the wipes is to bring them to the same temperature as the bath water and thus to prevent any factors arising from a temperature difference. Immediately the bathing procedure is commenced, a chronometer will be started by a nurse who is independent of the study.

After bathing, the patient's bedsheets and clothing will be changed and waste will be removed from the area. If the bandaging in the patient's operation area has not yet been removed, the operation area will not be washed. Also, the chronometer will be stopped by a nurse who is independent of the study immediately after the bathing procedure is completed, and the time taken for the procedure will be entered on the form.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over,
* Having upper and lower extremities,
* Good capillary filling,
* Systolic blood pressure is between 90-150 mmHg,
* SaO2 value of 90% and above,
* Willing to participate in the research

Exclusion Criteria:

* Serious burns and/or diarrhea
* Open wound bandaging or amputations of the upper or lower extremities
* Discharged or die during data collection
* Do not agree to participate in the study will not be included in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 5 months
  heart rate in minute

SECONDARY OUTCOMES:
Secondary Outcome Measure | 5 months
  blood pressure in mmHg

OTHER OUTCOMES:
Third Outcome Measure | 5 months
  body temperature in degrees celsius
Fourth Outcome Measure | 5 months
  breathing rate in minute
Fifth Outcome Measure | 5 months
  oxygen saturation values in percent
Sixth Outcome Measure | 5 months
  time taken for bathing in minute
Seventh Outcome Measure | 5 months
  weight in kilograms
Eighth Outcome Measure | 5 months
  height in meters
Ninth Outcome Measure | 5 months
  BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Şenay Yiğit Avcı, MSc, Study Chair — General Surgery Intensive Care Unit of Bursa Uludağ University Health Applications Research Center
Locations (1):
- Bursa Uludağ University, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toledo LV, Salgado PO, Souza CC, Brinati LM, Januario CF, Ercole FF. Effects of dry and traditional bed bathing on respiratory parameters: a randomized pilot study. Rev Lat Am Enfermagem. 2020;28:e3264. doi: 10.1590/1518-8345.3668.3264. Epub 2020 Jun 1. PMID 32491124
- [Background] Larson EL, Ciliberti T, Chantler C, Abraham J, Lazaro EM, Venturanza M, Pancholi P. Comparison of traditional and disposable bed baths in critically ill patients. Am J Crit Care. 2004 May;13(3):235-41. PMID 15149058
- [Background] Groven FMV, Zwakhalen SMG, Odekerken-Schroder G, Tan F, Hamers JPH. Comfort during the bed bath-A randomised crossover trial on the effect of washing without water versus water and soap in nursing students. J Clin Nurs. 2021 Aug;30(15-16):2234-2245. doi: 10.1111/jocn.15610. Epub 2021 May 6. PMID 33352004